CLINICAL TRIAL: NCT05324917
Title: Population Pharmacokinetic-pharmacodynamic Study of Rituximab in Children With Blood Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: YQ-KY-202101
Record Dates: First submitted 2022-02-28; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Rituximab; Children; Blood Disease
MeSH Terms: conditions — Hematologic Diseases | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lymphoma patients: Patients with Burkitt's lymphoma, diffuse large B-cell lymphoma, follicular lymphoma and other mature B-lymphoma patients. Patients were randomly divided into two groups for PK blood collection. There were 12 blood sampling sites in each group.
  Interventions: Drug: Rituximab
- Patients with B lymphoproliferative diseases: Patients with hematopoietic stem cell transplantation and Epstein-Barr virus associated b-cell lymphoproliferative diseases, b-cell lymphoproliferative changes, immune thrombocytopenia, and autoimmune hemolytic anemia. Patients were randomly divided into two groups for pharmacokinetics blood collection. There were 12 blood sampling sites in each group.
  Interventions: Drug: Rituximab (once a week)

INTERVENTIONS:
Drug: Rituximab — Chemotherapy for children with lymphoma: rituximab (375mg/m2 BSA) was added intravenously from COPADM1 regimen. once every 3 weeks to 4 weeks, combined with corresponding chemotherapy, a total of 4 times.
  Other Names: Rituximab injection
  Groups: lymphoma patients
Drug: Rituximab (once a week) — Rituximab (375mg/m2 BSA) was administered intravenously for lymphoproliferative diseases and EB virus-associated B lymphoproliferative diseases after hematopoietic stem cell transplantation. Once a week, a total of 4 times.
  ITP and AIHA patients received rituximab (100mg/m2 BSA) intravenously once a week, a total of 4 times.
  Other Names: Rituximab injection (once a week)
  Groups: Patients with B lymphoproliferative diseases

SUMMARY:
To establish a population pharmacokinetic and pharmacodynamic model of rituximab in children with hemopathy. To optimize the administration of rituximab in the treatment of children based on pharmacokinetic model.

DETAILED DESCRIPTION:
hemotherapy for children with lymphoma: rituximab (375mg/m2 BSA) was added intravenously from COPADM1 regimen. once every 3 weeks to 4 weeks, combined with corresponding chemotherapy, a total of 4 times.

Rituximab (375mg/m2 BSA) was administered intravenously for lymphoproliferative diseases and Epstein-Barr(EB) virus-associated B lymphoproliferative diseases after hematopoietic stem cell transplantation. Once a week, a total of 4 times.

Primary immunologic thrombocytopenic purpura(ITP) and autoimmune hemolytic anemia(AIAH) patients received rituximab (100mg/m2 BSA) intravenously once a week, a total of 4 times.

The children were divided into group A and group B according to the disease type, and each group was randomly divided into two groups (group 1 and group 2) and assigned blood collection points.

Burkitt's lymphoma diffuse large B-cell lymphoma follicular lymphoma and other mature B-lymphomas were in group A. Hematopoietic stem cell transplantation, EPstein-Barr virus associated lymphocyte proliferative disease, lymphocyte proliferative change, primary immunologic thrombocytopenic purpura(ITP) and autoimmune hemolytic anemia(AIAH) were in group B.

Group 1: Children in the first group were collected 0, 12, 24, and 72 h after the first dose, 0h before and after the second dose, 0h before and after the third dose, 0h before and after the last dose, 48, and 96 h after the last dose. Venous blood was collected at 12 time points.

Group 2: Children in the second group were collected 0, 12, 48, and 96 h after the first dose, 0h before and after the second dose, 0h before and after the third dose, 0h before and after the last dose, 24, and 72 h after the last dose. Venous blood was collected at 12 time points.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 18 years (including 6 months and 18 years), male or female.
* Burkitt's lymphoma, diffuse large B-cell lymphoma, follicular lymphoma and other mature B-cell lymphoma confirmed by histology or cytology, hematopoietic stem cell transplantation, EB virus associated B-cell proliferative diseases, b-cell proliferative changes, immune thrombocytopenia, Autoimmune hemolytic anemia and other patients with rituximab indications should be treated with rituximab monotherapy or combination.
* Eastern Cooperative Oncology Group(ECOG) physical status score was 0-2.
* Life expectancy was at least six months.
* Women and men with reproductive potential must agree to use effective contraceptive methods during and after treatment.
* The subjects or their parents or guardians fully know and sign the informed consent, and the subjects can cooperate to complete the follow-up.

Exclusion Criteria:

* Patients with known hypersensitivity to rituximab and rat protein.
* Previously known active infection of human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV), except for the following patients: Hepatitis B infection [hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb) positive] but negative results of HBV DNA polymerase chain reaction (PCR) can be included in the group.
* A confirmed history of progressive multifocal leukoencephalopathy (PML).
* Exclusion criteria associated with rituximab: tumor cell CD20 negative.
* Received live vaccine within 4 weeks prior to enrollment.
* Received immunoglobulin therapy within 3 months prior to enrollment.
* Participants in the clinical trials of other drugs and taking the test drugs within 3 months.
* Any other medical condition, metabolic abnormality, physical abnormality, or laboratory abnormality of clinical significance that, in the investigator's judgment, has reason to suspect that the patient has a medical condition or condition unsuitable for rituximab or that would affect the interpretation of study results or place the patient at high risk.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Age 6 months to 18 years, histologically or cytologically proven mature B lymphoma such as Burkitt's lymphoma, diffuse large B cell lymphoma, follicular lymphoma, hematopoietic stem cell transplantation, and Epstein-Barr virus associated B lymphoproliferative disease, B cell lymphoproliferative alteration, immune thrombocytopenia. Children with autoimmune hemolytic anemia and other diseases that meet the indication of rituximab and need rituximab monotherapy or combination therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-10 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
concentration of rituximab in plasma | 400 days
  the data of plasma drug concentration and time.

SECONDARY OUTCOMES:
Incidence of adverse events | 400 days
  Adverse events were recorded to evaluate the safety of the studied drugs.

IPD SHARING:
Plan to Share IPD: No